CLINICAL TRIAL: NCT04757038
Title: An Open Label, Randomized-controlled Trial to Assess Efficacy and Safety of HYALODISC Combined With Physical Exercise Program (PEP) Compared to Standard Care PEP in Patients With Low Back Pain Due to Degenerative Disc Disease
Brief Title: An Open Label, Randomized-controlled Trial to Assess Efficacy Safety of HYALODISC With Physical Exercise Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fidia Farmaceutici s.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EQM2.20.01
Record Dates: First submitted 2021-02-10; First posted 2021-02-16 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Degenerative Disc Disease(DDD)
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyalodisc injection (Experimental): • Group 1: One single X-ray-guided intradiscal injection (25 gauge) of 8 mg/mL of HYALODISC combined with PEP. The investigator will use one syringe for each involved disc, up to a maximum of three discs.
  The injection will be administered at V1 baseline (day 0). Any physical activity (e.g. jogging, tennis, weightlifting, prolonged upright position) in the 48 hours following the injection should be avoided. Both groups (Group 1 and Group 2) will be treated with PEP according to a standardized protocol.
  Interventions: Device: Intradiscal injection
- Physical exercise program (PEP) (No Intervention): Group 2: PEP alone

INTERVENTIONS:
Device: Intradiscal injection — The injection will be administered at V1 baseline (day 0). Any physical activity (e.g. jogging, tennis, weightlifting, prolonged upright position) in the 48 hours following the injection should be avoided.
  Other Names: Hyalodisc Injection
  Arms: Hyalodisc injection

SUMMARY:
The objective of this study is to determine if one single X-ray-guided intradiscal injection of 8 mg/mL of HYALODISC combined with PEP will be more effective than only physical exercise program in patients with LBP from degenerative disc disease.

Enrolled patients will be randomly assigned to one of the two treatment groups below:

* Group 1: One single X-ray-guided intradiscal injection (25 gauge) of 8 mg/mL of HYALODISC combined with PEP. The investigator will use one syringe for each involved disc, up to a maximum of three discs.
* Group 2: PEP alone. The injection will be administered at V1 baseline (day 0). Any physical activity (e.g. jogging, tennis, weightlifting, prolonged upright position) in the 48 hours following the injection should be avoided.

Both groups (Group 1 and Group 2) will be treated with PEP according to a standardized protocol. Starting one week after the baseline visit (V1), patients will be prescribed of 18 physiotherapy sessions that will take place under supervision of physiotherapist twice a week in the first seven weeks (weeks 2-8) and once a week in the next four weeks (weeks 9-12). Twelve repetitions of each exercise for 3 sets will be performed during PEP session. Moreover, in addition to the 18 sessions performed with supervision of the physiotherapist, all patients will be instructed how to do exercises at home and will be asked to continue these exercises once a week in the first seven weeks (weeks 2-8) and twice a week in the next four weeks (weeks 9-12).

DETAILED DESCRIPTION:
During the inclusion visit (V0) upon signature of the informed consent, eligible subject will be enrolled. At baseline visit (V1) eligible subjects will then randomly assigned to 1 of 2 treatment groups: HYALODISC + PEP (Group 1) or PEP alone (Group 2). At baseline visit (V1) HYALODISC (8 mg/ml) will be administered to group 1. The investigator will use one syringe for each involved disc, up to a maximum of three discs. The maximum volume that could be injected is 1.5 mL for each disc involved.

The PEP session will start for both groups one week after V1. Randomized subjects will follow the instructions during the PEP session, for a total of 18 sessions that will be performed under supervision of physiotherapist twice a week in the first seven weeks (weeks 2-8) and once a week in the next four weeks (weeks 9-12). Twelve repetitions of each exercise for 3 sets will be performed during PEP session. Moreover, all patients will be instructed how to continue these exercises at home, where the execution will be once a week in the first seven weeks (weeks 2-8) and twice a week in the next four weeks (weeks 9-12). Patients in group 2 that still present low back pain score > 6, despite the PEP, at the physical examination at V3 (12 weeks after V1), could be treated with HYALODISC intradiscally. Those patients will be then evaluated at 12 weeks after the treatment (week 24).

Follow-up visits are set at 4, 12 and 24 weeks (V2, V3 and V4)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18-70 years;
2. Written informed consent;
3. Willing and able to comply with the protocol for the duration of the study;
4. Chronic low back pain for at least 3 months from the screening;
5. Patients with at least one lumbar (L1-S1) black disc (Pfirrmann grade III-V) seen on magnetic resonance imaging (MRI) examination (MRI performed within 4 months from the screening visit);
6. Low back pain score of at least 5 on a 0-10 NRS at screening;
7. Roland-Morris Disability Questionnaire score of at least 9 on the 24-point questionnaire at screening;
8. If female of childbearing potential, must have a negative pregnancy test at screening and agree to use a reliable form of contraception throughout the study*.

Note: To be considered of non-childbearing potential, females must be surgically sterile or postmenopausal for at least 1 year.

* Highly effective birth control methods include: combined hormonal contraception (containing estrogen and progestogen) associated with inhibition of ovulation (oral, intravaginal, transdermal); progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable); intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; vasectomised partner; sexual abstinence..

Exclusion Criteria:

1. Cauda equina syndrome;
2. Active malignancy or tumours as source of symptoms;
3. Current infection or prior history of spinal infection (e.g., discitis, septic arthritis, epidural abscess) or an active systemic infection;
4. Previous lumbar spine surgery;
5. Evidence of prior lumbar vertebral body fracture;
6. Patients with radiculopathy caused by nerve root compression;
7. Verbiest Syndrome of Lumbar Spine;
8. Spondylolisthesis (> Grade 1) with or without spondylolysis at the symptomatic level(s);
9. Radiological sacroiliac joint involvement;
10. Patients with positive response to medial branch block;
11. Patients that did physical exercise therapy in the last three months before screening;
12. For patients that need to perform a MRI at the screening visit, contraindications to perform the MRI, such as patients carrying cerebral clips or cooling, valvular endoprosthesis with metal components, defibrillators, pacemakers or neurostimulant devices;
13. Sacrum-iliac synchondrosis agenesis seen on MRI;
14. Patients with symptomatic hernia, sciatica or spinal cord injury:
15. Significant systemic disease, including unstable angina, autoimmune disease, rheumatoid arthritis, and muscular dystrophy;
16. Congenital or acquired coagulopathy or thrombocytopenia; or currently taking anticoagulant, antineoplastic, antiplatelet, or thrombocytopenia-inducing medications; or undergoing radiation therapy;
17. Patients with known allergies, hypersensitivity or intolerance to paracetamol and/or active or inactive excipients of formulation;
18. Ongoing or previous participation in another drug or device clinical study within the previous 2 months from the screening;
19. Females known to be pregnant or nursing at time of enrolment or with plans to become pregnant within the planned length of follow-up or unwilling to use adequate contraception and conduct a pregnancy test at screening;
20. Patients with suspected or known history of hypersensitivity to hyaluronic acid or to hyaluronate preparations or gram-positive bacterial proteins;
21. Patients unable to provide a valid informed consent or those acting in an emergency situation..

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-07-02 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain reduction will be measured as difference of Numerical Rating Scale (NRS) value at Week 12 vs. baseline. The mean change in NRS score from baseline to Week 12 will be the primary efficacy endpoint. | week 12
  Pain reduction will be measured as difference of Numerical Rating Scale (NRS) value at Week 12 vs. baseline in terms of mean change in NRS score from baseline to Week 12 will be the primary efficacy endpoint

SECONDARY OUTCOMES:
To evaluate pain reduction, after treatment with HYALODISC + PEP compared to PEP alone; | week 4 and 24
  Pain reduction, measured as the mean change in NRS score from baseline to Week 4 and 24
To evaluate black disc hydration after HYALODISC + PEP, compared to PEP alone; | week 12 and 24
  Black disc hydration, measured as the percentage of patients with a reduction of at least one Pfirrmann grade.It will be evaluated by MRI at Week 12 and 24
To evaluate patient's response to therapy according Roland-Morris Disability Questionnaire (RMDQ) | week 4 ,12 and 24
  RMDQ, administered at screening and at week 4, 12 and 24 to evaluate clinical improvement after the treatment compared to the control group. The mean change in RMDQ score from baseline to Wee4, 12 and 24 will be considered for this endpoint
To evaluate quality of life assessed by the mean change from baseline in the EuroQol 5-Dimension Questionnaire, 5-level version (EQ-5D-5L) Index | week 12 and 24
  The mean change in EQ-5D-5L score from baseline to Week 12 and 24
To evaluate Patient's and investigator's global assessment of patient's health status (COGA/PTGA) | week 4, 12 and 24
  COGA /PTGA measured as the mean change in VAS (mm) from baseline to Week 4, Week 12, and Week 24
To evaluate Consumption of daily rescue medication (paracetamol) | week 4,12,24
  Rescue medications consumption, reported by the patient using a daily diary in which the usage of rescue medication (paracetamol) will be recorded as number of rescue medications taken for LBP. The diary will be evaluated at week 4, 12 and 24 after treatment and compared to the control group. The number of patients who take at least one dose of rescue medication as well as the total amount of rescue medication taken over the study will be analyzed
Consumption of daily rescue medication (paracetamol) | week 4,12,24
  Rescue medications consumption, reported by the patient using a daily diary in which the usage of rescue medication (paracetamol) will be recorded as rescue medications taken for LBP. The diary will be evaluated at week 4, 12 and 24 after treatment and compared to the control group. The percentage of patients who take at least one dose of rescue medication as well as the total amount of rescue medication taken over the study will be analyzed
To evaluate the safety profile and the local tolerability of HYALODISC. | through study completion
  Evaluated in terms of incidence of adverse events over the 24 weeks of the study.All adverse events (AEs) which occur during the study after the Subject has signed the ICF and (for Group 1) has received at least one dose of the product under investigation, whether referred by Subject, discovered by investigator questioning, or detected through physical examination, or by other means, must be collected and reported in the eCRF.
  As far as possible, each adverse event will be described by:
  * Duration (start and end dates);
  * Severity grade (mild, moderate, severe);
  * Causality (relationship) to the study product;
  * Action(s) taken;
  * Outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Marcia, Principal Investigator — Presidio Ospedaliero SS Trinità Cagliari; Eva Koetsier, Principal Investigator — Ospedale Regionale di Lugano
Locations (2):
- Unità operativa complessa di Radiologia PO.SS.Trinità, Cagliari, Italy
- Centro per la Terapia del Dolore NSI-EOC FMH Anestesiologia S.S.I.P.M.. Ospedale, Viganello, Lugano, Switzerland